CLINICAL TRIAL: NCT03991130
Title: High Dose IL-2 in Combination With Anti-PD-1 to Overcome Anti-PD-1 Resistance in Metastatic Melanoma and Renal Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Gregory Daniels (Other)
Responsible Party: Sponsor-Investigator, Gregory Daniels, Clinical Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCSD IIT HD IL-2; NCT03889782 (obsolete NCT alias)
Record Dates: First submitted 2019-06-16; First posted 2019-06-19 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Melanoma Stage Iv; Renal Cell Carcinoma, Metastatic
Keywords: melanoma; renal cell carcinoma
MeSH Terms: conditions — Melanoma; Carcinoma, Renal Cell; Neoplasm Metastasis | interventions — Interleukin-2; Nivolumab; spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- High Dose IL-2 and Nivolumab (Experimental)
  Interventions: Drug: IL-2 and Nivolumab

INTERVENTIONS:
Drug: IL-2 and Nivolumab — Course length will be 35 days. Subjects will receive 480 mg IV of nivolumab on day 1 of the cycle. The patient will be admitted to UCSD Jacobs Medical center for standard HD IL-2 which will be administered every 8 hrs for up to 14 doses days 8-12 per institutional practice. The patient will be readmitted days 22-28 for HD IL-2 every 8 hrs for up to 14 doses. Nivolumab 480 mg IV will be administered day 35. Scans for response will occur 4 weeks after day 35 nivolumab dose and response will be determined by RECIST 1.1 to determine if the patient will receive the next course.
  Other Names: High Dose IL-2; Anti-PD-1

SUMMARY:
The primary objective of this single arm phase 2 trial is to assess the response rate [complete response (CR) + partial response (PR)] of combined nivolumab and HD IL-2 in subjects with metastatic melanoma and renal cell carcinoma. Response will be performed after each course of nivolumab and IL-2 using RECIST 1.1. Patients will be treated for one course past best response for a maximum of 3 courses.

DETAILED DESCRIPTION:
PrimaryObjective Determine the overall response rate (complete response and partial response) for patients receiving anti-PD-1 (nivolumab) and high dose IL-2 (HD IL-2) in subjects with metastatic melanoma or renal cell carcinoma who have previously progressed on anti-PD-1 therapy. Response assessment will be performed using revised RECIST guideline (v 1.1).

Secondary Objectives

* Characterize safety, tolerability and adverse effects (AE) profile of nivolumab with HD IL-2 in subjects with metastatic malignant melanoma or renal cell carcinoma
* Measure Progression-Free Survival (PFS) using RECIST 1.1 after completion of at least one course of therapy (2 doses of nivolumab, 2 cycles of HD IL-2) for subjects enrolled in the study.

ExploratoryObjectives

* Correlate PD-L1 expression and tumor mutational burden (TMB) in archived diagnostic tumor tissue with best clinical response for subjects with metastatic melanoma and renal cell carcinoma
* Correlate myeloid-derived suppressor cells and T-cell subsets in peripheral blood during therapy with best clinical response (RECIST criteria) and treatment outcome in subjects with metastatic melanoma or renal cell carcinoma. Data will be collected prior to each treatment and after each course of treatment.

Study Duration: 48 months Amount of Subjects: up to 25 subjects

ELIGIBILITY:
Inclusion Criteria:

* Patient has the ability to understand and the willingness to sign a written informed consent.
* Age ≥ 18 years at the time of consent.
* At least 6 weeks of prior anti-PD-1 therapy with documented clinical or radiographic progression. Last anti-PD-1 therapy must be within 6 months of enrollment.
* Histologically-confirmed diagnosis of unresectable stage III or metastatic (stage IV) melanoma or renal cell carcinoma
* Measurable disease, defined as at least 1 tumor that fulfills the criteria for a target lesion according to RECIST 1.1, and obtained by imaging within 28 days prior registration for protocol therapy.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 28 days prior to registration for protocol therapy.
* Adequate hepatic function within 28 days prior to registration for protocol therapy defined as meeting all of the following criteria:
* total bilirubin ≤ 1.5 × upper limit of normal (ULN) OR direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 x ULN (except in patients with Gilbert's syndrome who must have a total bilirubin less than 3.0 mg/dl.)

  * and aspartate aminotransferase (AST) ≤ 2.5 × ULN or ≤ 5 × ULN for subjects with known hepatic metastases
  * and alanine aminotransferase (ALT) ≤ 2.5 × ULN or ≤ 5 × ULN for subjects with known hepatic metastases
* Adequate renal function within 28 days prior to registration for protocol therapy defined by either of the following criteria:

  * Serum creatinine ≤ 1.5 mg/dL
  * OR if serum creatinine > 1.5 mg/dL, estimated glomerular filtration rate (GFR) ≥ 50 mL/min
* Adequate hematologic function within 28 days prior to registration for protocol therapy defined as meeting all of the following criteria:

  * hemoglobin ≥ 9.0 g/dL
  * and absolute neutrophil count (ANC) ≥ 1000/L without the support of filgrastim
  * white blood cells (WBC) ≥ 3000/L
  * and platelet count ≥ 100 × 109/L
* Adequate coagulation functioning within 28 days prior to registration for protocol therapy defined by either of the following criteria:

  * INR < 1.5 × ULN
  * OR for subjects receiving warfarin or LMWH, the subjects must, in the investigator's opinion, be clinically stable with no evidence of active bleeding while receiving anticoagulant therapy. The INR for these subjects may exceed 1.5 × ULN if that is the goal of anticoagulant therapy.
* Adequate pulmonary and cardiac function for HD IL-2 (will be assessed clinically)
* Female subjects of childbearing potential must have confirmed negative urine or serum pregnancy test prior to drug administration and be willing to use two methods of birth control.
* Male subjects who are not surgically sterile (vasectomy) must agree to use an adequate method of contraception.
* Subject's toxicities from prior treatments must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo)

Exclusion Criteria:

* Active infection requiring systemic therapy
* Women who are pregnant or breastfeeding.
* Second active malignancy within the past 5 years with the exception of localized basal or squamous cell skin cancer, in situ cervical or bladder cancer, or localized prostate cancer under active surveillance.
* Active symptomatic central nervous system (CNS) metastases. Prior treated metastases or asymptomatic metastases are allowed. Patient can receive radiation between treatments if deemed medically necessary.
* Surgery within 4 weeks prior to study treatment except for minor procedures.
* Uncontrolled or poorly-controlled hypertension (> 160 mmHg systolic or > 100 mmHg diastolic for > 4 weeks) despite standard medical management.
* Serious or non-healing wounds, ulcers, or bone fractures within 28 days prior to initiation of study treatment.
* Any arterial thromboembolic events, including but not limited to myocardial infarction, transient ischemic attack, cerebrovascular accident, or unstable angina, within 6 months prior to initiation of study treatment.
* Has any condition that, in the opinion of the investigator, might jeopardize the safety of the patient or interfere with protocol compliance.
* Has any mental or medical condition that prevents the patient from giving informed consent or participating in the trial.
* Known hypersensitivity to nivolumab or IL-2 or any of their components.
* Known history of active tuberculosis.
* Concurrent systemic steroid therapy with doses above physiologic level (more than 10 mg of prednisone daily).
* Active autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with anti-phospholipid syndrome, granulomatosis with polyangiitis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis requiring treatment. Patients cannot be on immunosuppressive medications other than physiologic replacement doses of prednisone (less than 10 mg per day at enrollment) or equivalent steroid. Asymptomatic patients or those stable on non-immunosuppressive medications are eligible.
* Treatment with any investigational agent within 21 days prior to initiation of study treatment and the subject must have recovered from the acute toxic effects of the regimen with the exception of prior anti-PD-1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | 3 years post treatment
  The primary endpoint will be the response rate [complete response (CR) and partial response (PR)] of combined therapy with nivolumab and HD IL-2 in metastatic melanoma and renal cell carcinoma and will be evaluated using revised RECIST 1.1. Response rate will be computed with associated 95% confidence intervals.

SECONDARY OUTCOMES:
Drug Toxicity | After Initiation of a 35 day study treatment period up to 90 days following the last administration of study treatment
  Proportion of subjects with each grade of adverse events as defined by CTCAE v 5.0 will be computed. Toxicity will be reported in a tabular and descriptive manner.
Progression Free Survival | 1 year +/- 3 months
  • Median PFS times will be calculate and PFS rate at 1 year +/- 3 months will be calculated with associated 95% confidence intervals based on the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego Moores Cancer Center, La Jolla, California, United States